CLINICAL TRIAL: NCT05218850
Title: Butyrate Therapy in Hispanic Children With Ulcerative Colitis
Brief Title: The Use of Butyrate Therapy in Pediatric Ulcerative Colitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Sonia Michail, MD, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-22-00049; 161396 (Other: IND)
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Butyrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- open label intervention arm (Experimental): Butyrate enemas will be administered once daily for twelve weeks.
  Interventions: Drug: Butyrate

INTERVENTIONS:
Drug: Butyrate — Butyrate enemas will be administered once a day for 12 weeks
  Other Names: Butyrate enemas

SUMMARY:
Butyrate is an important metabolite produced by the gut microbiome and has been shown as a helpful therapy in ulcerative colitis. This is a feasibility study to determine the efficacy of butryate enemas in pediatric ulcerative colitis.

DETAILED DESCRIPTION:
butyrate enemas will be administered for 12 weeks to children ages 7 to 21 with mild to moderate ulcerative colitis to determine if butyrate therapy can help improve the clinical disease in those children. standard management of the disease will be performed during these 12 weeks including routine laboratory studies and endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* 7-21 years, mild to moderate ulcerative colitis

Exclusion Criteria:

* UC therapy within 4 weeks of study medication initiation
* infectious colitis, -pregnancy

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
remission of clinical disease | 12 weeks
  pediatric ulcerative colitis activity index, remission is <10, mild disease 10-34, moderate 35-64, severe 65 or greater

SECONDARY OUTCOMES:
improvement of inflammatory markers including ESR, CRP, Calprotectin | 12 weeks
  normalization or at least improvement of inflammatory markers described above

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Michail, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
data can be shared upon request